CLINICAL TRIAL: NCT01215188
Title: A Multicenter, Double-Blind Study of the Safety, Tolerability, and Immunogenicity of Pneumococcal Conjugate Vaccine (V114) Compared to Prevnar 13™ in Healthy Infants
Brief Title: A Study of Pneumococcal Conjugate Vaccine (V114) Compared to a Marketed Vaccine (V114-003)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: V114-003; V114-003 (Other: Merck Protocol Number)
Record Dates: First submitted 2010-10-04; First posted 2010-10-06 (Estimated); Results first posted 2019-04-30 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Pneumococcal Infections
Keywords: Invasive pneumococcal disease; Pneumonia; Pneumococcal conjugate vaccine
MeSH Terms: conditions — Pneumococcal Infections; Pneumonia | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- V114 Aluminum-adjuvanted (Experimental): Four intramuscular (IM) doses at 0.5 mL of aluminum-adjuvanted V114 pneumococcal conjugate vaccine at 2, 4, 6, and 12 to 15 months of age.
  Interventions: Biological: V114 Aluminum-adjuvanted
- V114 Non-adjuvanted (Experimental): Four IM doses at 0.5 mL of non-adjuvanted V114 pneumococcal conjugate vaccine at 2, 4, 6, and 12 to 15 months of age.
  Interventions: Biological: V114 Non-adjuvanted
- Prevnar 13® (Active Comparator): Four IM doses at 0.5 mL of Prevnar 13® at 2, 4, 6, and 12 to 15 months of age.
  Interventions: Biological: Prevnar 13®

INTERVENTIONS:
Biological: V114 Aluminum-adjuvanted — 15-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, 33F (2.2 mcg each), serotype 6B (4.4 mcg) and aluminum phosphate adjuvant (125 mcg) in each 0.5 mL dose.
  Arms: V114 Aluminum-adjuvanted
Biological: V114 Non-adjuvanted — 15-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, 33F (2 mcg each), and serotype 6B (4 mcg) in each 0.5 mL dose.
  Arms: V114 Non-adjuvanted
Biological: Prevnar 13® — 13-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 23F (2.2 mcg each), serotype 6B (4.4 mcg each) and aluminum phosphate adjuvant (125 mcg) in each 0.5. mL dose.
  Arms: Prevnar 13®

SUMMARY:
This study will evaluate whether the aluminum-adjuvanted or the non-adjuvanted formulation of the candidate pneumococcal vaccine (V114) is non-inferior to Prevnar 13® based on immune responses to the 13 serotypes in common Prevnar 13®

ELIGIBILITY:
Inclusion criteria:

* Healthy infants ≥ 42 days to ≤ 89 days.
* Participant's parent/legal guardian understands the study procedures, alternate treatments available and risks involved with the study, and voluntarily agrees to allow the child to participate by giving written informed consent.
* Afebrile, with a rectal temperature <38.1°C (<100.5°F) or axillary temperature <37.8°C (<100.0°F) on day of vaccination.
* Participant's parent/legal guardian is able to read, understand, and complete study questionnaires (i.e., the Vaccination Report Card).
* Participant is able to attend all scheduled visits and to comply with the study procedures.
* Participant's parent/legal guardian has access to a telephone.

Exclusion Criteria:

* Prior administration of any pneumococcal vaccine.
* Known hypersensitivity to any component of the pneumococcal conjugate vaccine.
* Known or suspected impairment of immunological function.
* Participant has a history of congenital or acquired immunodeficiency (e.g., splenomegaly).
* Participant or his/her mother has documented human immunodeficiency virus (HIV) infection.
* Functional or anatomic asplenia.
* History of autoimmune disease including multiple sclerosis (MS), systemic lupus, polymyositis, inclusion body myositis, dermatomyositis, Hashimoto's thyroiditis, Sjogren's syndrome, rheumatoid arthritis, other autoimmune disorders.
* Known neurologic or cognitive behavioral disorders including multiple sclerosis (MS), MS-like disease, encephalitis/myelitis, acute disseminating encephalomyelitis, pervasive developmental disorder, and related disorders.
* Use of any immunosuppressive therapy (Note: topical and inhaled/nebulized steroids are permitted). Participants on intramuscular, oral, or intravenous corticosteroid treatment should be excluded if they are receiving or expected to receive in the period from 30 days prior to Visit 1 through Visit 6 (30 days post-dose 4) more than 2 mg/kg per day of prednisone (or its equivalent), or more than 20 mg/d if they weigh more than 10 kg and are not otherwise immunocompromised. Excluded immunosuppressive therapies also include chemotherapeutic agents used to treat cancer or other conditions, and treatments associated with organ or bone marrow transplantation, or autoimmune disease.
* Participant has received other licensed non-live vaccines within the 14 days before receipt of study vaccine.
* Participant has received a licensed live virus vaccine within the 30 days prior of receipt of study vaccine.
* Prior receipt of a blood transfusion or blood products, including immunoglobulins.
* Investigational drugs or vaccines received within the 2 months before receipt of study vaccine.
* Participation in another clinical study within 42 days before the beginning or anytime during the duration of the current clinical study.
* History of invasive pneumococcal disease (positive blood culture, positive cerebrospinal fluid culture, or other sterile site) or known history of other culture positive pneumococcal disease.
* A recent febrile illness (rectal temperature ≥38.1°C [≥100.5°F]) occurring within 72 hours before receipt of study vaccine.
* History of failure to thrive.
* Participant has a coagulation disorder contraindicating IM vaccination.
* Participant and his/her mother have documented hepatitis B surface antigen-positive.
* Any infant who cannot be adequately followed for safety according to the protocol plan.
* Participant's parent/legal guardian is unlikely to adhere to study procedures, keep appointments, or is planning to relocate during the study.
* Any other reason that in the opinion of the investigator may interfere with the evaluation required by the study.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1152 (Actual)
Dates: Start 2010-10-14 (Actual); Primary Completion 2012-07-31 (Actual); Study Completion 2012-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Greenberg D, Hoover PA, Vesikari T, Peltier C, Hurley DC, McFetridge RD, Dallas M, Hartzel J, Marchese RD, Coller BG, Stek JE, Abeygunawardana C, Winters MA, MacNair JE, Pujar NS, Musey L. Safety and immunogenicity of 15-valent pneumococcal conjugate vaccine (PCV15) in healthy infants. Vaccine. 2018 Oct 29;36(45):6883-6891. doi: 10.1016/j.vaccine.2018.02.113. Epub 2018 Sep 21. PMID 30244873

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in 58 trial centers: 4 in Canada, 8 in Finland, 3 in Israel, 1 in Puerto Rico, 3 in Spain and 39 in the United States.
Pre-assignment Details: There were 1152 participants randomized into the study. The 1142 participants included in this study excluded 4 subjects who each received a combination of vaccines and who each had a final disposition of completed and excludes an additional 6 subjects who were randomized but never vaccinated.
Groups:
- V114 Adjuvanted: Participants received four intramuscular (IM) doses at 0.5 mL of aluminum-adjuvanted V114 pneumococcal conjugate vaccine at 2, 4, 6, and 12 to 15 months of age.
- V114 Nonadjuvanted: Participants received four IM doses at 0.5 mL of non-adjuvanted V114 pneumococcal conjugate vaccine at 2, 4, 6, and 12 to 15 months of age.
- PREVNAR 13®: Participants received four 0.5 mL IM doses of PREVNAR 13® at 2, 4, 6, and 12 to 15 months of age.
Period: Overall Study
Arm/Group | V114 Adjuvanted | V114 Nonadjuvanted | PREVNAR 13®
Started | 378 | 386 | 378
Completed | 320 | 327 | 326
Not Completed | 58 | 59 | 52
Not completed — Lost to Follow-up | 22 | 22 | 16
Not completed — Adverse Event | 1 | 1 | 3
Not completed — Physician Decision | 2 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 1 | 1
Not completed — Withdrawal by Subject | 32 | 34 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V114 Adjuvanted | V114 Nonadjuvanted | PREVNAR 13® | Total
Number analyzed (Participants) | 378 | 386 | 378 | 1142
Age, Customized [Mean (Standard Deviation); unit: Weeks] | 8.9 (1.2) | 8.8 (1.2) | 8.7 (1.1) | 8.8 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 177 | 189 | 179 | 545
  Male | 201 | 197 | 199 | 597
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 70 | 77 | 79 | 226
  Not Hispanic or Latino | 308 | 309 | 299 | 916
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 28 | 31 | 25 | 84
  Asian | 10 | 5 | 7 | 22
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 44 | 43 | 40 | 127
  White | 268 | 288 | 275 | 831
  More than one race | 27 | 18 | 31 | 76
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving the Immunoglobulin G (IgG) Serotype-specific ≥0.35 μg/mLThreshold Value for Postvaccination 3
Description: Percentage of participants meeting the serotype-specific IgG reference level (an antibody concentration measured by the pneumococcal polysaccharide electrochemiluminescence [Pn ECL] assay corresponding to the World Health Organization enzyme-linked immunosorbent assay [WHO ELISA] ≥ 0.35 μg/mL) (post-dose 3) for the 13 serotypes in common with PREVNAR 13® (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) and the 2 serotypes (serotypes 22F and 33F) not in common with PREVNAR 13®.
Time Frame: One month postvaccination 3
Population: The analysis population included all infant participants who did not have a protocol violation that could have impacted the validity of the antibody responses.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 Adjuvanted | V114 Nonadjuvanted | PREVNAR 13®
Number analyzed (Participants) | 300 | 315 | 315
Percentage of Participants
  Serotype 1 | 98.0 [95.7 to 99.3] | 96.2 [93.4 to 98.0] | 97.5 [95.1 to 98.9]
  Serotype 3 | 93.3 [89.9 to 95.9] | 89.8 [86.0 to 92.9] | 69.2 [63.8 to 74.3]
  Serotype 4 | 97.0 [94.4 to 98.6] | 94.0 [90.7 to 96.3] | 96.5 [93.8 to 98.2]
  Serotype 5 | 95.7 [92.7 to 97.7] | 92.4 [88.9 to 95.1] | 96.2 [93.4 to 98.0]
  Serotype 6A | 77.0 [71.8 to 81.6] | 78.4 [73.5 to 82.8] | 96.8 [94.2 to 98.5]
  Serotype 6B | 73.7 [68.3 to 78.6] | 65.4 [59.9 to 70.6] | 87.6 [83.5 to 91.0]
  Serotype 7F | 99.0 [97.1 to 100] | 99.4 [97.7 to 100] | 99.4 [97.7 to 100]
  Serotype 9V | 95.0 [91.9 to 97.2] | 92.4 [88.9 to 95.1] | 97.5 [95.1 to 98.9]
  Serotype 14 | 98.7 [96.6 to 100] | 98.4 [96.3 to 99.5] | 97.8 [95.5 to 99.1]
  Serotype 18C | 96.7 [94.0 to 98.4] | 89.8 [86.0 to 92.9] | 97.5 [95.1 to 98.9]
  Serotype 19A | 82.7 [77.9 to 86.8] | 84.4 [80.0 to 88.3] | 96.5 [93.8 to 98.2]
  Serotype 19F | 91.3 [87.6 to 94.3] | 91.1 [87.4 to 94.0] | 99.4 [97.7 to 100]
  Serotype 22F (non-PREVNAR 13® serotype) | 99.0 [97.1 to 100] | 99.4 [97.7 to 100] | 1.9 [0.7 to 4.1]
  Serotype 23F | 87.7 [83.4 to 91.2] | 81.6 [76.9 to 85.7] | 90.8 [87.0 to 93.7]
  Serotype 33F (non-PREVNAR 13® serotype) | 83.3 [78.6 to 87.4] | 84.8 [80.3 to 88.5] | 1.0 [0 to 2.8]

2. Primary Outcome: IgG Geometric Mean Concentrations (GMCs) for Postvaccination 3
Description: The IgG GMCs were evaluated as measured in the Pn ECL assay, for recipients of adjuvanted V114, non-adjuvanted V114, and Prevnar 13® (post-dose 3) for the 13 serotypes in common with PREVNAR 13® (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) and the 2 serotypes (serotypes 22F and 33F) not in common with PREVNAR 13®.
Time Frame: One month postvaccination 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | V114 Adjuvanted | V114 Nonadjuvanted | PREVNAR 13®
Number analyzed (Participants) | 300 | 315 | 315
µg/mL
  Serotype 1 | 1.34 [1.24 to 1.45] | 1.38 [1.27 to 1.51] | 1.84 [1.69 to 2.01]
  Serotype 3 | 0.95 [0.88 to 1.03] | 0.88 [0.81 to 0.96] | 0.50 [0.46 to 0.55]
  Serotype 4 | 1.28 [1.18 to 1.39] | 1.26 [1.16 to 1.37] | 1.32 [1.22 to 1.43]
  Serotype 5 | 1.61 [1.46 to 1.77] | 1.53 [1.38 to 1.71] | 1.83 [1.65 to 2.02]
  Serotype 6A | 0.93 [0.80 to 1.08] | 0.93 [0.80 to 1.07] | 2.91 [2.62 to 3.24]
  Serotype 6B | 0.95 [0.78 to 1.15] | 0.69 [0.57 to 0.84] | 1.47 [1.27 to 1.69]
  Serotype 7F | 2.63 [2.41 to 2.87] | 2.66 [2.44 to 2.90] | 3.67 [3.40 to 3.97]
  Serotype 9V | 1.49 [1.35 to 1.64] | 1.29 [1.16 to 1.44] | 1.79 [1.63 to 1.97]
  Serotype 14 | 4.17 [3.76 to 4.63] | 3.84 [3.43 to 4.29] | 5.62 [5.02 to 6.28]
  Serotype 18C | 1.27 [1.17 to 1.39] | 1.08 [0.97 to 1.20] | 1.99 [1.81 to 2.19]
  Serotype 19A | 0.90 [0.80 to 1.00] | 0.94 [0.84 to 1.05] | 2.05 [1.85 to 2.27]
  Serotype 19F | 1.50 [1.33 to 1.69] | 1.71 [1.52 to 1.93] | 2.54 [2.35 to 2.75]
  Serotype 22F (non-PREVNAR 13® serotype) | 5.24 [4.74 to 5.79] | 4.86 [4.40 to 5.37] | 0.07 [0.06 to 0.07]
  Serotype 23F | 1.05 [0.94 to 1.17] | 0.79 [0.69 to 0.89] | 1.41 [1.25 to 1.58]
  Serotype 33F (non-PREVNAR 13® serotype) | 1.47 [1.24 to 1.73] | 1.50 [1.29 to 1.74] | 0.06 [0.06 to 0.07]

3. Primary Outcome: IgG GMCs for Postvaccination 4
Description: The IgG GMCs were evaluated as measured in the Pn ECL assay, for recipients of adjuvanted V114, non-adjuvanted V114, and Prevnar 13® (post-dose 4) for the 13 serotypes in common with PREVNAR 13® (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) and the 2 serotypes (serotypes 22F and 33F) not in common with PREVNAR 13®.
Time Frame: One month postvaccination 4
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | V114 Adjuvanted | V114 Nonadjuvanted | PREVNAR 13®
Number analyzed (Participants) | 275 | 298 | 283
µg/mL
  Serotype 1 | 1.91 [1.73 to 2.10] | 1.81 [1.65 to 2.00] | 2.18 [1.99 to 2.38]
  Serotype 3: number analyzed (Participants) | 272 | 296 | 282
  Serotype 3 | 1.26 [1.15 to 1.39] | 1.12 [1.04 to 1.22] | 0.69 [0.63 to 0.75]
  Serotype 4: number analyzed (Participants) | 274 | 298 | 281
  Serotype 4 | 1.46 [1.30 to 1.65] | 1.40 [1.27 to 1.53] | 1.68 [1.52 to 1.86]
  Serotype 5: number analyzed (Participants) | 275 | 298 | 282
  Serotype 5 | 1.93 [1.74 to 2.14] | 1.79 [1.63 to 1.97] | 2.53 [2.28 to 2.81]
  Serotype 6A: number analyzed (Participants) | 274 | 297 | 279
  Serotype 6A | 3.78 [3.37 to 4.26] | 3.17 [2.81 to 3.57] | 6.55 [5.89 to 7.28]
  Serotype 6B: number analyzed (Participants) | 275 | 298 | 281
  Serotype 6B | 5.24 [4.68 to 5.86] | 3.98 [3.52 to 4.51] | 5.51 [4.90 to 6.20]
  Serotype 7F: number analyzed (Participants) | 274 | 298 | 282
  Serotype 7F | 4.18 [3.76 to 4.64] | 3.43 [3.14 to 3.75] | 5.73 [5.24 to 6.28]
  Serotype 9V: number analyzed (Participants) | 273 | 298 | 281
  Serotype 9V | 2.82 [2.52 to 3.15] | 2.50 [2.28 to 2.75] | 3.37 [3.04 to 3.72]
  Serotype 14: number analyzed (Participants) | 275 | 298 | 282
  Serotype 14 | 6.05 [5.37 to 6.82] | 5.55 [4.99 to 6.17] | 7.57 [6.81 to 8.42]
  Serotype 18C: number analyzed (Participants) | 275 | 298 | 281
  Serotype 18C | 2.14 [1.94 to 2.37] | 1.68 [1.54 to 1.83] | 3.37 [3.06 to 3.71]
  Serotype 19A: number analyzed (Participants) | 275 | 298 | 281
  Serotype 19A | 3.04 [2.72 to 3.40] | 3.42 [3.03 to 3.87] | 6.14 [5.57 to 6.78]
  Serotype 19F: number analyzed (Participants) | 275 | 298 | 282
  Serotype 19F | 5.56 [4.99 to 6.20] | 6.35 [5.68 to 7.09] | 4.51 [4.07 to 5.00]
  Serotype 22F (non-PREVNAR 13® serotype): number analyzed (Participants) | 272 | 298 | 283
  Serotype 22F (non-PREVNAR 13® serotype) | 9.64 [8.74 to 10.62] | 7.73 [7.08 to 8.45] | 0.12 [0.11 to 0.14]
  Serotype 23F: number analyzed (Participants) | 275 | 298 | 280
  Serotype 23F | 1.99 [1.75 to 2.26] | 1.61 [1.43 to 1.80] | 3.14 [2.78 to 3.54]
  Serotype 33F (non-PREVNAR 13® serotype): number analyzed (Participants) | 273 | 298 | 283
  Serotype 33F (non-PREVNAR 13® serotype) | 6.29 [5.62 to 7.05] | 4.95 [4.46 to 5.51] | 0.08 [0.08 to 0.09]

4. Primary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the Sponsor's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the Sponsor's product, is also an adverse experience.
Time Frame: Up to Day 14 postvaccination
Population: The analysis population included all randomized participants who received at least one dose of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | V114 Adjuvanted | V114 Nonadjuvanted | PREVNAR 13®
Number analyzed (Participants) | 368 | 382 | 376
Participants | 349 | 359 | 354

5. Primary Outcome: Number of Participants With an Injection-site AE
Description: Injection-site AEs reported by > 0% of participants in one or more vaccination groups were assessed.
Time Frame: Up to Day 14 postvaccination
Population: The analysis population included all randomized participants who received at least one dose of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | V114 Adjuvanted | V114 Nonadjuvanted | PREVNAR 13®
Number analyzed (Participants) | 368 | 382 | 376
Participants | 307 | 302 | 304

6. Primary Outcome: Number of Participants With a Systemic AE
Description: Systemic AEs reported by > 0% of participants in one or more vaccination groups were assessed.
Time Frame: Up to Day 14 postvaccination
Measure: Count of Participants; unit: Participants
Arm/Group | V114 Adjuvanted | V114 Nonadjuvanted | PREVNAR 13®
Number analyzed (Participants) | 368 | 382 | 376
Participants | 342 | 352 | 347

7. Primary Outcome: Number of Participants With a Serious Adverse Event (SAE)
Description: An SAE is an AE that results in death, is life threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment.
Time Frame: Up to one month after last dose of study vaccine
Population: The analysis population included all randomized participants who received at least one dose of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | V114 Adjuvanted | V114 Nonadjuvanted | PREVNAR 13®
Number analyzed (Participants) | 368 | 382 | 376
Participants | 25 | 27 | 29

8. Primary Outcome: Number of Participants Who Discontinued the Study Due to an AE
Description: as for outcome 4
Time Frame: Up to Day 14 postvaccination
Population: The analysis population included all randomized participants who received at least one dose of study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | V114 Adjuvanted | V114 Nonadjuvanted | PREVNAR 13®
Number analyzed (Participants) | 368 | 382 | 376
Participants | 1 | 1 | 2

9. Secondary Outcome: Percentage of Participants With Opsonophagocytic Killing Activity (OPA) Titer ≥ 8 as Measured by Fourfold Multiplexed Opsonization Assay (MOPA4) for Postvaccination 3
Description: The antibody responses as measured by MOPA4 (post-dose 3) for the 13 serotypes in common with PREVNAR 13® (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) and the 2 serotypes (serotypes 22F and 33F) not in common with PREVNAR 13®. Functional antibody activity was assessed only in a subset of the vaccinated participants, thus the study was not powered for assessing non-inferiority with respect to the OPA antibody responses.
Time Frame: One month postvaccination 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 Adjuvanted | V114 Nonadjuvanted | PREVNAR 13®
Number analyzed (Participants) | 120 | 120 | 122
Percentage of Participants
  Serotype 1: number analyzed (Participants) | 120 | 120 | 121
  Serotype 1 | 80.0 [71.7 to 86.7] | 73.3 [64.5 to 81.0] | 77.7 [69.2 to 84.8]
  Serotype 3 | 99.2 [95.4 to 100] | 100.0 [97.0 to 100] | 100.0 [97.0 to 100]
  Serotype 4: number analyzed (Participants) | 120 | 119 | 121
  Serotype 4 | 100.0 [97.0 to 100] | 100.0 [96.9 to 100] | 100.0 [97.0 to 100]
  Serotype 5 | 99.2 [95.4 to 100] | 95.8 [90.5 to 98.6] | 97.5 [93.0 to 99.5]
  Serotype 6A | 89.2 [82.2 to 94.1] | 85.8 [78.3 to 91.5] | 100.0 [97.0 to 100]
  Serotype 6B: number analyzed (Participants) | 119 | 120 | 121
  Serotype 6B | 84.0 [76.2 to 90.1] | 80.0 [71.7 to 86.7] | 96.7 [91.8 to 99.1]
  Serotype 7F | 100.0 [97.0 to 100] | 100.0 [97.0 to 100] | 100.0 [97.0 to 100]
  Serotype 9V: number analyzed (Participants) | 120 | 119 | 122
  Serotype 9V | 100.0 [97.0 to 100] | 98.3 [94.1 to 100] | 99.2 [95.5 to 100]
  Serotype 14 | 100.0 [97.0 to 100] | 99.2 [95.4 to 100] | 100.0 [97.0 to 100]
  Serotype 18C | 99.2 [95.4 to 100] | 96.7 [91.7 to 99.1] | 100.0 [97.0 to 100]
  Serotype 19A: number analyzed (Participants) | 120 | 119 | 122
  Serotype 19A | 92.5 [86.2 to 96.5] | 95.0 [89.3 to 98.1] | 95.9 [90.7 to 98.7]
  Serotype 19F | 95.0 [89.4 to 98.1] | 95.8 [90.5 to 98.6] | 99.2 [95.5 to 100]
  Serotype 22F (non-PREVNAR 13® serotype) | 99.2 [95.4 to 100] | 100.0 [97.0 to 100] | 11.6 [6.5 to 18.7]
  Serotype 23F: number analyzed (Participants) | 120 | 119 | 122
  Serotype 23F | 97.5 [92.9 to 99.5] | 96.6 [91.6 to 99.1] | 96.7 [91.8 to 99.1]
  Serotype 33F (non-PREVNAR 13® serotype) | 97.5 [92.9 to 99.5] | 99.2 [95.4 to 100] | 60.7 [51.4 to 69.4]

10. Secondary Outcome: Percentage of Participants With OPA Titer ≥ 8 as Measured by MOPA4 for Postvaccination 4
Description: The antibody responses as measured by MOPA4 (post-dose 4) for the 13 serotypes in common with PREVNAR 13® (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) and the 2 serotypes (serotypes 22F and 33F) not in common with PREVNAR 13®. Functional antibody activity was assessed only in a subset of the vaccinated participants, thus the study was not powered for assessing non-inferiority with respect to the OPA antibody responses.
Time Frame: One month postvaccination 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 Adjuvanted | V114 Nonadjuvanted | PREVNAR 13®
Number analyzed (Participants) | 58 | 59 | 50
Percentage of Participants
  Serotype 1 | 96.6 [88.1 to 100] | 94.9 [85.9 to 98.9] | 96.0 [86.3 to 100]
  Serotype 3 | 100.0 [93.8 to 100] | 100.0 [93.9 to 100] | 100.0 [92.9 to 100]
  Serotype 4 | 98.3 [90.8 to 100] | 100.0 [93.9 to 100] | 100.0 [92.9 to 100]
  Serotype 5 | 98.3 [90.8 to 100] | 100.0 [93.9 to 100] | 100.0 [92.9 to 100]
  Serotype 6A | 98.3 [90.8 to 100] | 100.0 [93.9 to 100] | 100.0 [92.9 to 100]
  Serotype 6B | 98.3 [90.8 to 100] | 100.0 [93.9 to 100] | 100.0 [92.9 to 100]
  Serotype 7F | 100.0 [93.8 to 100] | 100.0 [93.9 to 100] | 100.0 [92.9 to 100]
  Serotype 9V | 98.3 [90.8 to 100] | 100.0 [93.9 to 100] | 100.0 [92.9 to 100]
  Serotype 14 | 100.0 [93.8 to 100] | 100.0 [93.9 to 100] | 100.0 [92.9 to 100]
  Serotype 18C | 98.3 [90.8 to 100] | 100.0 [93.9 to 100] | 100.0 [92.9 to 100]
  Serotype 19A | 98.3 [90.8 to 100] | 98.3 [90.9 to 100] | 100.0 [92.9 to 100]
  Serotype 19F | 96.6 [88.1 to 100] | 100.0 [93.9 to 100] | 100.0 [92.9 to 100]
  Serotype 22F (non-PREVNAR 13® serotype) | 100.0 [93.8 to 100] | 100.0 [93.8 to 100] | 17.0 [7.6 to 30.8]
  Serotype 23F | 100.0 [93.8 to 100] | 100.0 [93.9 to 100] | 100.0 [92.9 to 100]
  Serotype 33F (non-PREVNAR 13® serotype) | 100.0 [93.8 to 100] | 100.0 [93.9 to 100] | 88.0 [75.7 to 95.5]

11. Secondary Outcome: OPA Geometric Mean Titers (GMTs) as Measured by MOPA4 for Postvaccination 3
Description: The antibody responses as measured by MOPA4 (post-dose 3) for the 13 serotypes in common with PREVNAR 13® (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) and the 2 serotypes (serotypes 22F and 33F) not in common with PREVNAR 13®. The OPA antibody responses included the percentage of participants with OPA titer and the GMTs. Functional antibody activity was assessed only in a subset of the vaccinated participants, thus the study was not powered for assessing non-inferiority with respect to the OPA antibody responses.
Time Frame: One month postvaccination 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114 Adjuvanted | V114 Nonadjuvanted | PREVNAR 13®
Number analyzed (Participants) | 120 | 120 | 122
μg/mL
  Serotype 1: number analyzed (Participants) | 120 | 120 | 121
  Serotype 1 | 35.4 [25.4 to 49.3] | 32.4 [22.5 to 46.5] | 44.6 [31.2 to 63.7]
  Serotype 3 | 296.7 [246.9 to 356.6] | 254.3 [215.9 to 299.6] | 209.9 [178.6 to 246.7]
  Serotype 4: number analyzed (Participants) | 120 | 119 | 121
  Serotype 4 | 1672.9 [1414.3 to 1978.7] | 1633.1 [1384.3 to 1926.6] | 1911.6 [1608.0 to 2272.4]
  Serotype 5: number analyzed (Participants) | 120 | 120 | 121
  Serotype 5 | 467.6 [369.4 to 591.7] | 337.0 [259.5 to 437.7] | 542.8 [416.8 to 706.7]
  Serotype 6A | 1273.6 [807.3 to 2009.1] | 703.3 [435.4 to 1136.1] | 4009.7 [3316.0 to 4848.4]
  Serotype 6B: number analyzed (Participants) | 119 | 120 | 121
  Serotype 6B | 765.5 [463.2 to 1265.2] | 419.5 [244.8 to 719.0] | 1597.5 [1145.7 to 2227.4]
  Serotype 7F | 5818.1 [4945.3 to 6844.8] | 5791.3 [4816.9 to 6962.9] | 10454.1 [8614.1 to 12687.0]
  Serotype 9V: number analyzed (Participants) | 120 | 119 | 122
  Serotype 9V | 2227.4 [1791.0 to 2770.1] | 1927.3 [1493.8 to 2486.5] | 2685.5 [2110.5 to 3417.1]
  Serotype 14 | 2266.2 [1835.9 to 2797.2] | 1574.8 [1232.4 to 2012.3] | 2786.5 [2244.3 to 3459.7]
  Serotype 18C | 1263.7 [1035.4 to 1542.2] | 846.6 [652.4 to 1098.8] | 2209.0 [1833.1 to 2662.0]
  Serotype 19A: number analyzed (Participants) | 120 | 119 | 122
  Serotype 19A | 551.7 [383.3 to 794.1] | 457.9 [331.1 to 633.3] | 1292.1 [921.9 to 1810.9]
  Serotype 19F | 986.2 [714.0 to 1362.2] | 933.7 [665.8 to 1309.5] | 1417.1 [1145.4 to 1753.3]
  Serotype 22F (non-PREVNAR 13® serotype): number analyzed (Participants) | 120 | 119 | 122
  Serotype 22F (non-PREVNAR 13® serotype) | 3048.8 [2484.3 to 3741.5] | 2714.4 [2302.6 to 3199.9] | 3.9 [2.8 to 5.5]
  Serotype 23F: number analyzed (Participants) | 120 | 119 | 122
  Serotype 23F | 1087.7 [821.8 to 1439.8] | 726.4 [530.3 to 995.1] | 3040.3 [2249.0 to 4110.1]
  Serotype 33F (non-PREVNAR 13® serotype) | 25075.2 [16645.2 to 37774.5] | 28262.3 [20745.0 to 38503.5] | 66.6 [39.0 to 113.7]

12. Secondary Outcome: OPA GMTs as Measured by MOPA4 for Postvaccination 4
Description: as for outcome 10
Time Frame: One month postvaccination 4
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114 Adjuvanted | V114 Nonadjuvanted | PREVNAR 13®
Number analyzed (Participants) | 58 | 59 | 50
μg/mL
  Serotype 1 | 139.1 [90.0 to 215.0] | 124.0 [79.6 to 192.9] | 133.1 [86.3 to 205.1]
  Serotype 3 | 438.6 [344.8 to 557.9] | 405.2 [330.0 to 497.4] | 369.7 [293.8 to 465.0]
  Serotype 4 | 1674.3 [1171.5 to 2392.9] | 1752.9 [1394.0 to 2204.0] | 2456.5 [1895.1 to 3184.2]
  Serotype 5 | 680.8 [474.7 to 976.6] | 866.5 [648.5 to 1157.9] | 830.3 [602.1 to 1144.8]
  Serotype 6A | 2583.6 [1667.0 to 4004.2] | 2835.9 [2171.6 to 3703.5] | 7382.0 [5445.2 to 10007.6]
  Serotype 6B | 3866.8 [2723.7 to 5489.7] | 2265.1 [1559.4 to 3290.2] | 4686.1 [3058.7 to 7179.3]
  Serotype 7F | 10205.9 [7487.6 to 13911.2] | 8543.2 [6622.6 to 11020.6] | 19147.5 [13725.9 to 26710.7]
  Serotype 9V | 2888.0 [1985.0 to 4201.7] | 3339.1 [2457.9 to 4536.2] | 4901.5 [3740.3 to 6423.2]
  Serotype 14 | 3543.1 [2508.3 to 5005.0] | 2877.7 [2088.7 to 3964.7] | 3872.9 [2762.1 to 5430.5]
  Serotype 18C | 1327.0 [945.3 to 1862.8] | 1171.1 [928.6 to 1476.9] | 3214.7 [2438.0 to 4238.9]
  Serotype 19A | 1871.0 [1282.1 to 2730.4] | 2260.8 [1604.8 to 3185.0] | 4519.7 [3028.7 to 6744.7]
  Serotype 19F | 1885.8 [1226.6 to 2899.2] | 2949.8 [2273.6 to 3827.0] | 2624.6 [1866.0 to 3691.5]
  Serotype 22F (non-PREVNAR 13® serotype) | 4586.5 [3406.2 to 6175.7] | 4497.0 [3594.5 to 5626.1] | 4.8 [2.6 to 8.8]
  Serotype 23F | 3118.0 [2203.2 to 4412.6] | 2469.2 [1904.5 to 3201.4] | 11490.0 [7815.4 to 16892.4]
  Serotype 33F (non-PREVNAR 13® serotype) | 59179.6 [43706.0 to 80131.4] | 54562.2 [38760.3 to 76806.2] | 815.8 [408.0 to 1631.3]

13. Secondary Outcome: Percentage of Participants Achieving the IgG Serotype-specific Threshold Value of ≥0.35 μg/mL for Postvaccination 4
Description: Percentage of participants achieving World Health Organization (WHO) predefined antibody threshold as measured by the pneumococcal polysaccharide electrochemiluminescence (Pn ECL) assay corresponding to the WHO enzyme-linked immunosorbent assay (ELISA) value of ≥ 0.35μg/mL (post-dose 4) for the 13 serotypes in common with PREVNAR 13® (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) and the 2 serotypes (serotypes 22F and 33F) not in common with PREVNAR 13®.
Time Frame: One month postvaccination 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 Adjuvanted | V114 Nonadjuvanted | PREVNAR 13®
Number analyzed (Participants) | 300 | 315 | 315
Percentage of Participants
  Serotype 1: number analyzed (Participants) | 275 | 298 | 283
  Serotype 1 | 98.2 [95.8 to 99.4] | 98.0 [95.7 to 99.3] | 100.0 [98.7 to 100]
  Serotype 3: number analyzed (Participants) | 272 | 296 | 282
  Serotype 3 | 96.0 [92.9 to 98.0] | 95.9 [93.0 to 97.9] | 80.9 [75.8 to 85.3]
  Serotype 4: number analyzed (Participants) | 274 | 298 | 281
  Serotype 4 | 95.6 [92.5 to 97.7] | 96.3 [93.5 to 98.1] | 96.8 [94.0 to 98.5]
  Serotype 5: number analyzed (Participants) | 275 | 298 | 282
  Serotype 5 | 99.3 [97.4 to 100] | 99.0 [97.1 to 100] | 98.9 [96.9 to 100]
  Serotype 6A: number analyzed (Participants) | 274 | 297 | 279
  Serotype 6A | 98.5 [96.3 to 100] | 97.3 [94.8 to 98.8] | 99.6 [98.0 to 100]
  Serotype 6B: number analyzed (Participants) | 275 | 298 | 281
  Serotype 6B | 99.3 [97.4 to 100] | 97.7 [95.2 to 99.1] | 98.9 [96.9 to 100]
  Serotype 7F: number analyzed (Participants) | 274 | 298 | 282
  Serotype 7F | 100.0 [98.7 to 100] | 99.0 [97.1 to 100] | 99.6 [98.0 to 100]
  Serotype 9V: number analyzed (Participants) | 273 | 298 | 281
  Serotype 9V | 98.9 [96.8 to 100] | 99.0 [97.1 to 100] | 99.6 [98.0 to 100]
  Serotype 14: number analyzed (Participants) | 275 | 298 | 282
  Serotype 14 | 99.6 [98.0 to 100] | 99.7 [98.1 to 100] | 100.0 [98.7 to 100]
  Serotype 18C: number analyzed (Participants) | 275 | 298 | 281
  Serotype 18C | 98.5 [96.3 to 100] | 99.0 [97.1 to 100] | 100.0 [98.7 to 100]
  Serotype 19A: number analyzed (Participants) | 275 | 298 | 281
  Serotype 19A | 97.5 [94.8 to 99.0] | 98.7 [96.6 to 100] | 100.0 [98.7 to 100]
  Serotype 19F: number analyzed (Participants) | 275 | 298 | 282
  Serotype 19F | 99.3 [97.4 to 100] | 99.0 [97.1 to 100] | 99.3 [97.5 to 100]
  Serotype 22F (non-PREVNAR 13® serotype): number analyzed (Participants) | 272 | 298 | 283
  Serotype 22F (non-PREVNAR 13® serotype) | 100.0 [98.7 to 100] | 99.7 [98.1 to 100] | 7.4 [4.7 to 11.1]
  Serotype 23F: number analyzed (Participants) | 275 | 298 | 280
  Serotype 23F | 95.6 [92.5 to 97.7] | 95.0 [91.8 to 97.2] | 98.9 [96.9 to 100]
  Serotype 33F (non-PREVNAR 13® serotype): number analyzed (Participants) | 273 | 298 | 283
  Serotype 33F (non-PREVNAR 13® serotype) | 98.9 [96.8 to 100] | 98.3 [96.1 to 99.5] | 4.9 [2.7 to 8.2]

14. Secondary Outcome: Percentage of Participants Achieving the IgG Serotype-specific Threshold Value of ≥1.0 μg/mL for Postvaccination 4
Description: Percentage of participants achieving WHO predefined antibody threshold as measured by the Pn ECL assay corresponding to the WHO enzyme-linked immunosorbent assay (ELISA) value of ≥ 1.0 μg/mL (post-dose 4) for the 13 serotypes in common with PREVNAR 13® (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) and the 2 serotypes (serotypes 22F and 33F) not in common with PREVNAR 13®.
Time Frame: One month postvaccination 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 Adjuvanted | V114 Nonadjuvanted | PREVNAR 13®
Number analyzed (Participants) | 275 | 298 | 283
Percentage of Participants
  Serotype 1 | 77.5 [72.1 to 82.3] | 76.5 [71.3 to 81.2] | 84.1 [79.3 to 88.2]
  Serotype 3: number analyzed (Participants) | 272 | 296 | 282
  Serotype 3 | 63.6 [57.6 to 69.3] | 56.8 [50.9 to 62.5] | 30.9 [25.5 to 36.6]
  Serotype 4: number analyzed (Participants) | 274 | 298 | 281
  Serotype 4 | 62.0 [56.0 to 67.8] | 65.1 [59.4 to 70.5] | 73.3 [67.7 to 78.4]
  Serotype 5: number analyzed (Participants) | 275 | 298 | 282
  Serotype 5 | 79.6 [74.4 to 84.2] | 75.8 [70.6 to 80.6] | 85.1 [80.4 to 89.1]
  Serotype 6A: number analyzed (Participants) | 274 | 297 | 279
  Serotype 6A | 89.8 [85.6 to 93.1] | 89.2 [85.1 to 92.5] | 97.5 [94.9 to 99.0]
  Serotype 6B: number analyzed (Participants) | 275 | 298 | 281
  Serotype 6B | 97.1 [94.3 to 98.7] | 92.6 [89.0 to 95.3] | 95.4 [92.2 to 97.5]
  Serotype 7F: number analyzed (Participants) | 274 | 298 | 282
  Serotype 7F | 96.4 [93.4 to 98.2] | 97.0 [94.3 to 98.6] | 99.3 [97.5 to 100]
  Serotype 9V: number analyzed (Participants) | 273 | 298 | 281
  Serotype 9V | 88.6 [84.3 to 92.2] | 87.9 [83.7 to 91.4] | 91.5 [87.6 to 94.5]
  Serotype 14: number analyzed (Participants) | 275 | 298 | 282
  Serotype 14 | 95.3 [92.1 to 97.5] | 97.0 [94.3 to 98.6] | 98.2 [95.9 to 99.4]
  Serotype 18C: number analyzed (Participants) | 275 | 298 | 281
  Serotype 18C | 83.6 [78.7 to 87.8] | 74.5 [69.2 to 79.3] | 95.0 [91.8 to 97.2]
  Serotype 19A: number analyzed (Participants) | 275 | 298 | 281
  Serotype 19A | 87.6 [83.2 to 91.3] | 87.9 [83.7 to 91.4] | 96.4 [93.6 to 98.3]
  Serotype 19F: number analyzed (Participants) | 275 | 298 | 282
  Serotype 19F | 95.3 [92.1 to 97.5] | 97.0 [94.3 to 98.6] | 95.7 [92.7 to 97.8]
  Serotype 22F (non-PREVNAR 13® serotype): number analyzed (Participants) | 272 | 298 | 283
  Serotype 22F (non-PREVNAR 13® serotype) | 99.6 [98.0 to 100] | 98.7 [96.6 to 100] | 2.8 [1.2 to 5.5]
  Serotype 23F: number analyzed (Participants) | 275 | 298 | 280
  Serotype 23F | 76.4 [70.9 to 81.3] | 70.5 [64.9 to 75.6] | 86.4 [81.9 to 90.2]
  Serotype 33F (non-PREVNAR 13® serotype): number analyzed (Participants) | 273 | 298 | 283
  Serotype 33F (non-PREVNAR 13® serotype) | 96.0 [92.9 to 98.0] | 96.6 [93.9 to 98.4] | 1.4 [0 to 3.6]

ADVERSE EVENTS:
Time Frame: Up to 1 month after final vaccination
Description: The safety population consisted of all randomized participants who received study vaccine.
Groups:
- V114: Participants received four intramuscular (IM) doses at 0.5 mL of aluminum-adjuvanted V114 pneumococcal conjugate vaccine at 2, 4, 6, and 12 to 15 months of age.
- V114 Non-Adjuvanted: Participants received four IM doses at 0.5 mL of non-adjuvanted V114 pneumococcal conjugate vaccine at 2, 4, 6, and 12 to 15 months of age.
- Prevnar: Participants received four 0.5 mL IM doses of PREVNAR 13® at 2, 4, 6, and 12 to 15 months of age.
Arm/Group | V114 | V114 Non-Adjuvanted | Prevnar
All-Cause Mortality (participants affected / at risk) | 1/368 | 1/382 | 2/376
Serious Adverse Events (participants affected / at risk) | 25/368 | 27/382 | 29/376
Other Adverse Events (participants affected / at risk) | 345/368 | 348/382 | 347/376
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=368) | V114 Non-Adjuvanted (N=382) | Prevnar (N=376)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Developmental delay (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Sudden infant death syndrome (General disorders) | 1 (1) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 5 (5) | 6 (6) | 4 (5)
Bronchitis (Infections and infestations) | 0 (0) | 2 (4) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 3 (3)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastritis viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (4) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Lobar pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 2 (3)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 6 (6) | 7 (7) | 6 (6)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Unresponsive to stimuli (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Breath holding (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=368) | V114 Non-Adjuvanted (N=382) | Prevnar (N=376)
Constipation (Gastrointestinal disorders) | 19 (19) | 3 (3) | 14 (15)
Diarrhoea (Gastrointestinal disorders) | 36 (38) | 26 (29) | 36 (39)
Vomiting (Gastrointestinal disorders) | 17 (20) | 25 (28) | 25 (27)
Injection site erythema (General disorders) | 217 (475) | 179 (348) | 201 (400)
Injection site induration (General disorders) | 163 (314) | 112 (180) | 160 (324)
Injection site pain (General disorders) | 264 (687) | 280 (632) | 271 (647)
Injection site swelling (General disorders) | 181 (378) | 132 (235) | 165 (332)
Irritability (General disorders) | 315 (1072) | 311 (1005) | 306 (988)
Pyrexia (General disorders) | 123 (197) | 86 (147) | 110 (186)
Nasopharyngitis (Infections and infestations) | 22 (22) | 22 (27) | 21 (22)
Otitis media (Infections and infestations) | 29 (29) | 28 (28) | 22 (23)
Upper respiratory tract infection (Infections and infestations) | 30 (32) | 41 (44) | 26 (32)
Decreased appetite (Metabolism and nutrition disorders) | 212 (492) | 195 (405) | 196 (397)
Somnolence (Nervous system disorders) | 263 (743) | 281 (756) | 265 (689)
Cough (Respiratory, thoracic and mediastinal disorders) | 28 (30) | 25 (28) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.